CLINICAL TRIAL: NCT05400642
Title: SctO2 Evaluated by NIRS Between Apneic Oxygenation With High-flow Oxygen Therapy and Tracheal Intubation During Laryngeal Microsurgery: a Prospective Non-inferiority RCT
Brief Title: Randomized Controlled Trial:High-flow Oxygen Therapy and Tracheal Intubation for Laryngeal Microsurgery
Acronym: NIRS_ORL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4953
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Laryngeal Disease
Keywords: general anesthesia; hfnco; NIRS
MeSH Terms: conditions — Laryngeal Diseases | interventions — Tobacco Use Cessation Devices; Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Oxygen Therapy (Experimental): Surgery conducted under High Flow Oxygen Therapy
  Interventions: Device: THRIVE
- Mechanical ventilation (Active Comparator): Surgery conducted under orotracheal intubation and mechanical ventilation
  Interventions: Device: mechanical ventilation

INTERVENTIONS:
Device: THRIVE — Apneic ventilation
  Arms: High Flow Oxygen Therapy
Device: mechanical ventilation — mechanical ventilation in Positive Pressure
  Arms: Mechanical ventilation

SUMMARY:
Over time, the accumulation of carbon dioxide reduces the pressure gradient for the alveolar transfer of oxygen, limiting the successful duration of apneic oxygenation. NIRS (Near-Infrared Spectroscopy) technology is able to provide an estimate of the regional balance between demand and supply of brain oxygen.

The primary hypothesis of this study is that although high-flow oxygen therapy may be associated with transiently higher PaCO2 values than those found in patients undergoing tracheal intubation and traditional mechanical ventilation, due to the brevity of this phenomenon the variations in the average values of frontal cerebral tissue oxygen saturation are expected to be of similar magnitude between the two groups.

Secondary objectives will be the comparison of the success rate of high-flow oxygen therapy compared to traditional airway management by mechanical ventilation.

The success rate will be defined as blood pressure of carbon dioxide (PaCO2) <= 65 mmHg and/or peripheral oxygen saturation (SpO2) >= 94% throughout the procedure, in the absence of adverse events (haemodynamic alteration, dyspnea, discomfort).

The data will be analyzed according to an intention-to-treat principle. Continuous variables with repeated measurements will be compared with a mixed-effect linear regression model. Normality of distribution will be verified with the Shapiro-Wilk test. Continuous variables will be compared with Student t- or Mann-Whitney test; categorical variables with the Chi-square test.

DETAILED DESCRIPTION:
Apneic oxygenation is a physiological phenomenon in which, provided that patency exists between the lungs and the external environment, the pulmonary flow of oxygen is maintained by a negative pressure gradient generated by the difference between the rate of alveolar extraction of oxygen and the excretion of carbon dioxide.

Over time, the accumulation of carbon dioxide reduces the pressure gradient for the alveolar transfer of oxygen, limiting, because of a condition of acidosis, the successful duration of apneic oxygenation.

The effects of hypercapnia on the mechanisms of cerebral blood flow autoregulation are well known and NIRS (Near-Infrared Spectroscopy) technology, through the non-invasive analysis of the relative absorbance of oxy- and deoxyhemoglobin in the frontal cerebral tissue microcirculation, is able to provide an estimate of the regional balance between demand and supply of brain oxygen.

High-Flow Nasal Cannula Oxygenation (HFNCO) is an open-loop oxygenation system that uses flows of up to 70 l/min of 100% oxygen through the Optiflow THRIVETM apparatus (Fisher and Paykel Healthcare Ltd, Auckland, New Zealand), increasingly used as an alternative to tracheal intubation in patients undergoing short-term general anesthesia.

Heating and humidification of the flows facilitate their tolerability by the patient; HFNCO produces a linear, flow-dependent effect of continuous positive airway pressure about 1 cmH20 for every 10 l/min increase in oxygen flows, reduces dead space and allows elimination of carbon dioxide, with the potential to increase alveolar volume and improve gas exchanges.

The efficacy of HFNCO in apneic patients undergoing laryngeal surgery is debated: on the one hand it allows minimal manipulation of the airways by the anesthesiologist, it expands the surgical field and it proved to be not inferior to tracheal intubation in maintaining oxygen saturation, however it has been associated with a higher incidence of hypercapnia and the need for rescue maneuvers of airway management.

Laryngeal microsurgery includes procedures usually lasting < 30 minutes, performed under general anesthesia and tracheal intubation.

The primary hypothesis of this study is that although high-flow oxygen therapy may be associated with transiently higher PaCO2 values than those found in patients undergoing tracheal intubation and traditional mechanical ventilation, due to the brevity of this phenomenon the variations in the average values of frontal cerebral tissue oxygen saturation are expected to be of similar magnitude between the two groups.

Secondary objectives will be the comparison of the success rate of high-flow oxygen therapy compared to traditional airway management by mechanical ventilation.

The success rate will be defined as blood pressure of carbon dioxide (PaCO2) <= 65 mmHg and/or peripheral oxygen saturation (SpO2) >= 94% throughout the procedure, in the absence of adverse events.

The maximum arterial concentration of carbon dioxide achieved during the procedure, the percentage of complications in terms of inability to manage the airways with the need for tracheal intubation in the group treated with high-flow oxygen therapy, episodes of hypotension, cardiac arrhythmias and post-operative nausea and vomiting will also be compared; finally, the degree of dyspnea (with the Borg dyspnea score) and patient comfort (Visual Analogue Scale) at the end of the procedure will be evaluated.

The data will be analyzed according to an intention-to-treat principle. Clinical and demographic characteristics of the sample will be described through descriptive statistical techniques. Continuous quantitative variables with normal distribution will be reported as mean and standard deviation; as median and interquartile range the non-normal variables.

The confidence intervals for median differences will be calculated by the Hodges-Lehman method.

Categorical variables and missing data will be presented as absolute value and percentage, n (%). Continuous variables will be compared with the Student t-test in case of normal distribution or, if not, with the Mann-Whitney test for independent samples. The normality of the distribution of the variables will be verified graphically by histograms and with the Shapiro-Wilk test.

Differences between categorical variables will be analyzed using the Chi-square test or the Fisher's exact test in case of expected frequencies < 5.

For each participant, for SctO2, a combined average will be calculated (SctO2 left + SctO2 right/2).

Continuous variables with repeated measurements will be compared with a mixed-effect linear regression model, with correction according to Bonferroni's method. The type of airway management used and the timing at which the measurements will be performed will be considered as fixed effects; a random effect related to the patient will also be added.

ELIGIBILITY:
Inclusion Criteria:

ASA I and II. Scheduled for Microlaryngeal surgery

Exclusion Criteria:

1. age < 18 years;
2. pregnancy status;
3. NYHA class > III;
4. BMI > 30;
5. pre-existing cardiac arrhythmias;
6. high risk of inhalation;
7. neuromuscular diseases or metabolite accumulation;
8. refusal of informed consent or impossibility to express it.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
NIRS | each five minutes from anesthesia induction up to the end of surgery
  Average values of frontal cerebral tissue oxygen saturation

SECONDARY OUTCOMES:
The success rate of high-flow oxygen therapy compared to traditional airway management by mechanical ventilation. | each five minutes from anesthesia induction up to the end of surgery
  The success rate will be defined as blood pressure of carbon dioxide (PaCO2) <= 65 mmHg and/or peripheral oxygen saturation (SpO2) >= 94% throughout the procedure, in the absence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: fabio sbaraglia, phD, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fabio Sbaraglia, Roma, Italy

IPD SHARING:
Plan to Share IPD: No